CLINICAL TRIAL: NCT04198766
Title: An Open-Label, Multicenter, First-in-Human, Dose-Escalation, Multicohort, Phase 1/2 Study of INBRX-106 and INBRX-106 in Combination With Pembrolizumab in Subjects With Locally Advanced or Metastatic Solid Tumors
Brief Title: Study of INBRX-106 and INBRX-106 in Combination With Pembrolizumab (Keytruda®) in Subjects With Locally Advanced or Metastatic Solid Tumors (Hexavalent OX40 Agonist)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Inhibrx Biosciences, Inc (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Ph 1 Ph 2 INBRX-106; KEYNOTE A99 and MK-3475-A99 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor; Non-Small Cell Lung Cancer; Head and Neck Cancer; Melanoma; Gastric Cancer; Renal Cell Carcinoma; Urothelial Carcinoma
Keywords: Phase 1 and Phase 2; Phase 1 and Phase 2 Clinical Trial; Solid Tumors; Head and Neck Cancer; Lung Cancer; Non-Small Cell Lung Cancer; OX40 receptor agonist; PD-L1 positive; Pembrolizumab; Keytruda; Chemotherapy; Immunotherapy; HNSCC; Oropharyngeal cancer; Hypopharyngeal cancer; Oral cancer; INBRX-106; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Neoplasms; Neoplasms, Squamous Cell; Head and Neck Neoplasms; Neoplasms by Site; Carcinoma; Carcinoma, Squamous Cell; Molecular Mechanisms of Pharmacological Action; Antineoplastic Agents, Immunological; Antineoplastic Agents; Squamous Cell Carcinoma of Head and Neck; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Head and Neck Neoplasms; Melanoma; Stomach Neoplasms; Carcinoma, Renal Cell; Carcinoma, Transitional Cell; Lung Neoplasms; Squamous Cell Carcinoma of Head and Neck; Oropharyngeal Neoplasms; Hypopharyngeal Neoplasms; Mouth Neoplasms; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Neoplasms; Neoplasms, Squamous Cell; Neoplasms by Site; Carcinoma; Carcinoma, Squamous Cell | interventions — pembrolizumab; Pemetrexed; Cisplatin; Paclitaxel; Taxes

STUDY DESIGN:
Masking Description: Part 4 NSCLC cohort is randomized 1;1:1, open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- Part 1 INBRX-106 Escalation (Not Recruiting) (Experimental): INBRX-106 will be escalated in subjects with locally advanced or metastatic solid tumors.
  Interventions: Drug: INBRX-106 - Hexavalent OX40 agonist antibody
- Part 3 INBRX-106 Escalation in Combination with pembrolizumab (Not Recruiting) (Experimental): INBRX-106 will be escalated, in combination with pembrolizumab, in subjects with locally advanced or metastatic solid tumors.
  Interventions: Drug: INBRX-106 - Hexavalent OX40 agonist antibody; Drug: pembrolizumab 200 mg
- Part 2 (Cohorts C1/C2) INBRX-106 Escalation in Various Solid Tumor Types (Not Recruiting) (Experimental): Subjects with melanoma (any type), head and neck squamous cell carcinoma, renal cell carcinoma, urothelial carcinoma or MSI/TMB-high tumors that are relapsed or refractory to prior checkpoint inhibitor (CPI) therapy will be treated with INBRX-106
  Interventions: Drug: INBRX-106 - Hexavalent OX40 agonist antibody; Drug: pembrolizumab 200 mg
- Part 2 (Cohort C3) INBRX-106 Escalation in NSCLC (Not Recruiting) (Experimental): Subjects with non-small cell carcinoma relapsed or refractory to prior checkpoint inhibitor (CPI) therapy will be treated with INBRX-106
  Interventions: Drug: pembrolizumab 200 mg
- Part 4 (Cohort F3a) INBRX-106 Expansion in Combination with pembrolizumab in NSCLC (Not Recruiting) (Experimental): Subjects with non-small cell lung cancer will be treated with alternating dosing of INBRX-106 0.3 mg/kg Q6W and 400 mg pembrolizumab IV Q6W. This is one of the randomized cohorts.
  Interventions: Drug: INBRX-106 - Hexavalent OX40 agonist antibody; Drug: pembrolizumab 400 mg
- Part 4 (Cohort F3b) INBRX-106 Expansion in Combination with pembrolizumab in NSCLC (Not Recruiting) (Experimental): Subjects with non-small cell lung cancer will be given a 0.3 mg/kg priming dose of INBRX-106 in cycle 1, followed by 0.1 mg/kg INBRX-106 and 200 mg pembrolizumab IV every 3 weeks in subsequent cycles. This is one of the randomized cohorts.
  Interventions: Drug: INBRX-106 - Hexavalent OX40 agonist antibody; Drug: pembrolizumab 200 mg; Drug: pembrolizumab 400 mg
- Part 4 (Cohort F3c) Pembrolizumab Expansion Arm (Not Recruiting) (Active Comparator): Subjects with non-small cell lung cancer will be treated with 200 mg pembrolizumab IV every 3 weeks. This is one of the randomized cohorts.
  Interventions: Drug: INBRX-106 - Hexavalent OX40 agonist antibody
- Part 4 (Cohort F3d) INBRX-106 Expansion in Combination with pembrolizumab in NSCLC (concurrent) (Experimental): Subjects with non-small cell lung cancer will be treated concurrently every 6 weeks with INBRX-106 0.1 mg/kg and 200 mg pembrolizumab IV every 3 weeks. This is one of the randomized cohorts.
  Interventions: Drug: INBRX-106 - Hexavalent OX40 agonist antibody
- Part 4 (Cohort F4) INBRX-106 Expansion in Combination with pembrolizumab (Experimental): Subjects with melanoma (any type), head and neck squamous cell carcinoma (non-nasopharyngeal) OR nasopharyngeal carcinoma, MSI-high, TMB-high or MMR-deficient tumors, will be treated with INBRX-106 in combination with 200mg pembrolizumab IV every 3 weeks. Only NPC is currently enrolling.
  Interventions: Drug: INBRX-106 - Hexavalent OX40 agonist antibody; Drug: pembrolizumab 200 mg
- Part 4 (Cohort F5)INBRX-106 Expansion with pembrolizumab in MSI/TMB-high/MMRd tumors Not Recuriting (Experimental): Subjects with solid tumors that have confirmed MSI-high, TMB-high or MMR-deficient states who are relapsed or refractory to checkpoint inhibitor (CPI) therapy will be treated with INBRX-106 and 200 mg pembrolizumab IV every 3 weeks
  Interventions: Drug: INBRX-106 - Hexavalent OX40 agonist antibody; Drug: pembrolizumab 200 mg
- Part 4 (Cohort F6) INBRX-106 Expansion with pembrolizumab in Uveal Melanoma (Not Recruiting) (Experimental): Subjects with ocular (uveal) melanoma who are relapsed or refractory to checkpoint inhibitor (CPI) therapy will be treated with INBRX-106 and 200 mg pembrolizumab IV every 3 weeks
  Interventions: Drug: INBRX-106 - Hexavalent OX40 agonist antibody; Drug: pembrolizumab 200 mg; Drug: Carboplatin AUC-5; Drug: Pemetrexed 500 mg/m2
- Part 4 (Cohort F7a) INBRX-106 Expansion with pembrolizumab, pemetrexed and carboplatin in NSCLC (Experimental): This Arm is no longer recruiting. Subjects with advanced/metastatic NSCLC, any PD-L1 TPS will be treated with INBRX-106 0.1mg/kg, 200mg pembrolizumab, 500mg/m2 pemetrexed and carboplatin AUC-5 IV every 3 weeks
  Interventions: Drug: INBRX-106 - Hexavalent OX40 agonist antibody; Drug: pembrolizumab 200 mg; Drug: Pemetrexed 500 mg/m2; Drug: Cisplatin 75mg/m2
- Part 4 (Cohort F7b) INBRX-106 Expansion with pembrolizumab, pemetrexed and cisplatin in NSCLC (Experimental): This Arm is no longer recruiting. Subjects with advanced/metastatic NSCLC, any PD-L1 TPS will be treated with INBRX-106 0.1mg/kg, 200mg pembrolizumab, 500mg/m2 pemetrexed and 75mg/m2 cisplatin IV every 3 weeks
  Interventions: Drug: INBRX-106 - Hexavalent OX40 agonist antibody; Drug: pembrolizumab 200 mg; Drug: Carboplatin AUC-6; Drug: Paclitaxel 200mg/m2; Drug: Nab paclitaxel 100mg/m2
- Part 4(Cohort F7c)INBRX-106 Expansion with pembrolizumab, (Nab)-paclitaxel and carboplatin in NSCLC (Experimental): This Arm is no longer recruiting. Subjects with advanced/metastatic NSCLC, any PD-L1 TPS will be treated with INBRX-106 0.1mg/kg, 200mg pembrolizumab, 200mg/m2 paclitaxel and carboplatin AUC-6 IV every 3 weeks OR INBRX-106, 200mg pembrolizumab, 100mg/m2 nab-paclitaxel (dosed Days 1,8 and 15 every cycle) and carboplatin AUC-6 IV every 3 weeks. Treating physician to determine if paclitaxel or nab-paclitaxel will be given
  Interventions: Drug: INBRX-106 - Hexavalent OX40 agonist antibody; Drug: pembrolizumab 200 mg

INTERVENTIONS:
Drug: INBRX-106 - Hexavalent OX40 agonist antibody — The active ingredient of INBRX-106 is a recombinant, humanized, hexavalent IgG antibody that targets the human OX40 receptor (TNFRSF4).
  Arms: Part 1 INBRX-106 Escalation (Not Recruiting); Part 2 (Cohorts C1/C2) INBRX-106 Escalation in Various Solid Tumor Types (Not Recruiting); Part 3 INBRX-106 Escalation in Combination with pembrolizumab (Not Recruiting); Part 4 (Cohort F3a) INBRX-106 Expansion in Combination with pembrolizumab in NSCLC (Not Recruiting); Part 4 (Cohort F3b) INBRX-106 Expansion in Combination with pembrolizumab in NSCLC (Not Recruiting); Part 4 (Cohort F3c) Pembrolizumab Expansion Arm (Not Recruiting); Part 4 (Cohort F3d) INBRX-106 Expansion in Combination with pembrolizumab in NSCLC (concurrent); Part 4 (Cohort F4) INBRX-106 Expansion in Combination with pembrolizumab; Part 4 (Cohort F5)INBRX-106 Expansion with pembrolizumab in MSI/TMB-high/MMRd tumors Not Recuriting; Part 4 (Cohort F6) INBRX-106 Expansion with pembrolizumab in Uveal Melanoma (Not Recruiting); Part 4 (Cohort F7a) INBRX-106 Expansion with pembrolizumab, pemetrexed and carboplatin in NSCLC; Part 4 (Cohort F7b) INBRX-106 Expansion with pembrolizumab, pemetrexed and cisplatin in NSCLC; Part 4(Cohort F7c)INBRX-106 Expansion with pembrolizumab, (Nab)-paclitaxel and carboplatin in NSCLC
Drug: pembrolizumab 200 mg — pembrolizumab 200 mg by intravenous (IV) infusion, given on Day 1 of each 21-day cycle.
  Other Names: KEYTRUDA
  Arms: Part 2 (Cohort C3) INBRX-106 Escalation in NSCLC (Not Recruiting); Part 2 (Cohorts C1/C2) INBRX-106 Escalation in Various Solid Tumor Types (Not Recruiting); Part 3 INBRX-106 Escalation in Combination with pembrolizumab (Not Recruiting); Part 4 (Cohort F3b) INBRX-106 Expansion in Combination with pembrolizumab in NSCLC (Not Recruiting); Part 4 (Cohort F4) INBRX-106 Expansion in Combination with pembrolizumab; Part 4 (Cohort F5)INBRX-106 Expansion with pembrolizumab in MSI/TMB-high/MMRd tumors Not Recuriting; Part 4 (Cohort F6) INBRX-106 Expansion with pembrolizumab in Uveal Melanoma (Not Recruiting); Part 4 (Cohort F7a) INBRX-106 Expansion with pembrolizumab, pemetrexed and carboplatin in NSCLC; Part 4 (Cohort F7b) INBRX-106 Expansion with pembrolizumab, pemetrexed and cisplatin in NSCLC; Part 4(Cohort F7c)INBRX-106 Expansion with pembrolizumab, (Nab)-paclitaxel and carboplatin in NSCLC
Drug: pembrolizumab 400 mg — pembrolizumab 400 mg by IV infusion given on Day 1 of alternating 21-day cycles (every 6 weeks)
  Other Names: KEYTRUDA
  Arms: Part 4 (Cohort F3a) INBRX-106 Expansion in Combination with pembrolizumab in NSCLC (Not Recruiting); Part 4 (Cohort F3b) INBRX-106 Expansion in Combination with pembrolizumab in NSCLC (Not Recruiting)
Drug: Carboplatin AUC-5 — carboplatin AUC-5 by intravenous (IV) infusion, given on Day 1 of each 21-day cycle of cycles 1-4
  Arms: Part 4 (Cohort F6) INBRX-106 Expansion with pembrolizumab in Uveal Melanoma (Not Recruiting)
Drug: Carboplatin AUC-6 — carboplatin AUC-6 by intravenous (IV) infusion, given on Day 1 of each 21-day cycle of cycles 1-4
  Arms: Part 4 (Cohort F7b) INBRX-106 Expansion with pembrolizumab, pemetrexed and cisplatin in NSCLC
Drug: Pemetrexed 500 mg/m2 — pemetrexed 500 mg/m2 by IV infusion given on Day 1 of each 21-Day cycle for up to 35 cycles
  Other Names: Alimta®
  Arms: Part 4 (Cohort F6) INBRX-106 Expansion with pembrolizumab in Uveal Melanoma (Not Recruiting); Part 4 (Cohort F7a) INBRX-106 Expansion with pembrolizumab, pemetrexed and carboplatin in NSCLC
Drug: Cisplatin 75mg/m2 — cisplatin 75mg/m2 by intravenous (IV) infusion, given on Day 1 of each 21-day cycle of cycles 1-4
  Arms: Part 4 (Cohort F7a) INBRX-106 Expansion with pembrolizumab, pemetrexed and carboplatin in NSCLC
Drug: Paclitaxel 200mg/m2 — paclitaxel 200mg/m2 by intravenous (IV) infusion, given on Day 1 of each 21-day cycle of cycles 1-4
  Arms: Part 4 (Cohort F7b) INBRX-106 Expansion with pembrolizumab, pemetrexed and cisplatin in NSCLC
Drug: Nab paclitaxel 100mg/m2 — Nab paclitaxel 100mg/m2 by intravenous (IV) infusion, given on Days 1, 8 and 15 of each 21-day cycle of cycles 1-4
  Arms: Part 4 (Cohort F7b) INBRX-106 Expansion with pembrolizumab, pemetrexed and cisplatin in NSCLC

SUMMARY:
This is a Phase 1/2, open-label, non-randomized, 4-part trial to determine the safety profile and identify the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of INBRX 106 administered as a single agent or in combination with the anti-PD-1 checkpoint inhibitor (CPI) pembrolizumab (Keytruda®). KEYTRUDA is a registered trademark of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc., Rahway, NJ, USA.

ELIGIBILITY:
Select Inclusion Criteria:

* Males or females aged ≥18 years.
* Parts 1 and 3 (escalation cohorts): Subjects with locally advanced or metastatic non resectable solid tumors, whose disease has progressed despite all standard therapies or for whom no further standard or clinically acceptable therapy exists.
* Part 2 (single-agent expansion cohort): Subjects with NSCLC, melanoma, HNSCC, G/GEA, RCC, or TCC, with histologically confirmed, locally advanced or metastatic, non-resectable disease, which has progressed despite all standard therapies including CPI or for whom no standard or clinically acceptable therapy exists.
* Part 4 (expansion cohorts in combination with pembrolizumab, with or without chemotherapy): Subjects with melanoma (all types), HNSCC, G/GEA, RCC, TCC, NSCLC, or MSI-high, TMB-high, MMR-deficient tumors, with histologically confirmed, locally advanced or metastatic, non resectable disease, which is either CPI-naive (melanoma, HNSCC, NPC) or progressed despite all standard therapies including CPI (NSCLC, RCC, TCC, uveal melanoma, MSI-high, TMB-high, or MMR-deficient solid tumors) or for whom no standard or clinically acceptable therapy exists.
* For Cohort F3 (NSCLC), subjects may have progressed on no more than 2 lines of standard therapy that must include at least one PD-1/L1 regimen.
* For Cohort F4 (HNSCC and NPC), subjects may be previously treated with no more than 1 prior chemotherapy regimen in metastatic setting. Prior PD-1/L1 in curative (neo-adjuvant/adjuvant) setting is allowed only if completed >/= 6 months prior to progression to local recurrence or metastatic disease.
* All subjects with non-squamous NSCLC must have documentation of absence of tumor activating EGFR mutations and absence of ALK gene rearrangements.
* PD-L1 by IHC (22C3): Parts 1 and 3: IHC optional. Part 2: IHC result mandatory but any score allowed. Combined Positive Score (CPS) ≥ 1% (or Tumor Proportion Score ≥50% for NSCLC; for TMB-high tumors, any TPS% is allowed). Part 4: Combined Positive Score (CPS) ≥ 1% (or Tumor Proportion Score ≥50% for NSCLC; for TMB-high tumors, any TPS% is allowed).
* Adequate hematologic, coagulation, hepatic and renal function and ECOG score as defined per protocol.

Select Exclusion Criteria:

* Prior exposure to OX40 agonists.
* Receipt of any investigational product or any approved anticancer drug(s) or biological product(s) within 4 weeks prior to the first dose of study drug with certain exceptions.
* Hematologic malignancies (e.g., ALL, AML, MDS, CLL, CML, NHL, Hodgkin's lymphoma and multiple myeloma)
* Prior or concurrent malignancies. Exception: Subjects with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessments of INBRX-106.
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Exception: Subjects who are previously treated and are radiologically and clinically stable without the requirement for steroid treatment for at least 14 days prior to first dose of study treatment may be allowed study entry if certain criteria apply.
* Grade ≥ 3 immune-related adverse events (irAEs) or irAE that lead to discontinuation of prior immunotherapy. Some exceptions as defined per protocol apply.
* Active autoimmune disease or documented history of autoimmune disease that required systemic steroids or other immunosuppressive medications. Certain exceptions as defined in protocol apply.
* Diagnosis of immunodeficiency or treatment with systemic immunosuppressive medications within 7 days prior to the first dose of study drug. Certain exceptions as defined in protocol apply.
* History of hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) infection. Exceptions as defined in protocol apply.
* Active interstitial lung disease (ILD) or pneumonitis or a history of ILD or pneumonitis requiring treatment with steroids or other immunosuppressive medications.
* Clinically significant cardiac condition, including myocardial infarction, uncontrolled angina, cerebrovascular accident, or other acute uncontrolled heart disease < 3 months; left ventricular ejection fraction (LVEF) < 50%; New York Heart Association (NYHA) Class III or IV congestive heart failure; or uncontrolled hypertension; or oxygen saturation <92% on room air.
* Active, hemodynamically significant pulmonary embolism within 3 months prior to enrollment on this trial.
* Major surgery within 4 weeks prior to enrollment on this trial.
* Anti-infectious drug treatments (i.e., antibiotics) within 4 weeks prior to the first dose of study drug.
* Prior organ allograft transplantations or allogeneic peripheral blood stem cell (PBSC) or bone marrow (BM) transplantation.
* Additional in- and exclusion criteria per protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-05-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of adverse events of INBRX-106 as single agent and in combination with pembrolizumab | ~2 years
  Adverse events will be assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0
Severity of adverse events of INBRX-106 as single agent and in combination with pembrolizumab | ~2 years
  Adverse events will be assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0
MTD and/or RP2D of INBRX-106 as single agent and in combination with pembrolizumab | ~2 years
  Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D) of INBRX-106 and INBRX-106 in combination with pembrolizumab
Antitumor activity of INBRX-106 in combination with pembrolizumab in expansion cohorts | ~2 years
  Tumor response will be determined by immune Response Evaluation Criteria in Solid Tumors (iRECIST).
Frequency and severity of adverse events of INBRX-106 in combination with pembrolizumab and chemotherapy in adults with locally advanced or metastatic NSCLC | ~2 years
  Adverse events will be assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0

SECONDARY OUTCOMES:
Area under the serum concentration time curve (AUC) of INBRX-106 | ~2 years
  Area under the serum concentration time curve (AUC) of INBRX-106 as a single agent and in combination with pembrolizumab with or without chemotherapy will be determined.
Maximum observed serum concentration (Cmax) of INBRX-106 | ~2 years
  Maximum observed serum concentration (Cmax) of INBRX-106 as a single agent and in combination with pembrolizumab with or without chemotherapy will be determined.
Trough observed serum concentration (Ctrough) of INBRX-106 | ~2 years
  Trough observed serum concentration (Ctrough) of INBRX-106 as a single agent and in combination with pembrolizumab with or without chemotherapy will be determined.
Time to Cmax (Tmax) of INBRX-106 | ~2 years
  Time to Cmax (Tmax) of INBRX-106 as a single agent and in combination with pembrolizumab with or without chemotherapy will be determined.
Immunogenicity of INBRX-106 | ~2 years
  Frequency of anti-drug antibodies (ADA) against INBRX-106 as a single agent and in combination with pembrolizumab with or without chemotherapy will be determined.

OTHER OUTCOMES:
Anti-tumor activity of INBRX-106 as single agent and in combination with pembrolizumab with or without chemotherapy | ~2 years
  Tumor response will be determined by the revised Response Evaluation Criteria in Solid Tumors version 1.1 (RECISTv1.1).
Anti-tumor activity of INBRX-106 as single agent and in combination with pembrolizumab with or without chemotherapy | ~2 years
  Tumor response will be determined by immune Response Evaluation Criteria in Solid Tumors (iRECIST).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Lead, Study Director — Inhibrx Biosciences, Inc
Locations (42):
- United States (30):
  - City of Hope, Duarte, California
  - Los Angeles Cancer Network, Glendale, California
  - California Research Institute, Los Angeles, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - Valkyrie Clinical Trials, Murrieta, California
  - Providence Medical Foundation, Santa Rosa, California
  - Clermont Oncology Center, Clermont, Florida
  - Mid Florida Hematology and Oncology Center, Orange City, Florida
  - Winship Cancer Institute - Emory University, Atlanta, Georgia
  - The University of Chicago Medical Center, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Norton Cancer Institute, Louisville, Kentucky
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Cancer Institute, Detroit, Michigan
  - START Midwest, Grand Rapids, Michigan
  - HealthPartners Cancer Research Center, Saint Louis Park, Minnesota
  - HealthPartners Cancer Research Center (Regions Hospital), Saint Paul, Minnesota
  - Intermountain Health Cancer Centers of Montana, Billings, Montana
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Montefiore Medical Center, The Bronx, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Vanderbilt University School of Medicine, Nashville, Tennessee
  - Sarah Cannon Research Institute at Mary Crowley, Dallas, Texas
  - Renovatio Clinical - El Paso, El Paso, Texas
  - NEXT Oncology, San Antonio, Texas
  - Renovatio Clinical, The Woodlands, Texas
  - The University of Texas Health Science Center at Tyler, Tyler, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin
- Singapore (3):
  - Curie Oncology, Singapore
  - Icon Cancer Centre Farrer Park, Singapore
  - Icon Cancer Centre Mount Alvernia, Singapore
- South Korea (4):
  - The Catholic University of Korea, St. Vincent's Hospital, Gyeonggi-do
  - Asan Medical Center, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital,, Seoul
- Taiwan (5):
  - Changhua Christian Hospital (CCH), Changhua
  - E-Da Cancer Hospital, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital (KMUH), Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holay N, Yadav R, Ahn SJ, Kasiewicz MJ, Polovina A, Rolig AS, Staebler T, Becklund B, Simons ND, Koguchi Y, Eckelman BP, de Durana YD, Redmond WL. INBRX-106: a hexavalent OX40 agonist that drives superior antitumor responses via optimized receptor clustering. J Immunother Cancer. 2025 May 21;13(5):e011524. doi: 10.1136/jitc-2025-011524. PMID 40404202